CLINICAL TRIAL: NCT02564133
Title: Are Postoperative Complications More Frequent When Patients Having a Hip Fracture Have a Patent Foramen Ovale ?
Brief Title: Hip Fracture and Patent Foramen Ovale
Acronym: COL-FOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have discovered a too low prevalence of Patent Foramen Ovale compared to the theoretical % of around 20-25%.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/35; 2012-A01155-38 (Other: ANSM)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- detection of a patent foramen ovale (Experimental)
  Interventions: Device: Transthoracic echocardiography

INTERVENTIONS:
Device: Transthoracic echocardiography — A transthoracic echocardiography is performed to discover a patent foramen ovale

SUMMARY:
Ereth et al. showed in 1992, using transesophageal echocardiography, that the implantation of a hip prosthesis may be complicated by intracardiac embolization of various origin.

A patent foramen ovale exists in approximately one fifth of the population; it facilitates the passage of embolus from the right heart to the left one and then especially to the coronary vessels and to the brain.

The hypothesis supported in this research is that the prevalence of postoperative complications, especially neurological ones, is increased after surgery for hip fracture when patients have a patent foramen ovale.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture requiring a surgical procedure

Exclusion Criteria:

* simultaneous other traumatic lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative complications probably related to the presence of a patent foramen ovale | First postoperative week
  Complications probably related to the presence of a patent foramen ovale

SECONDARY OUTCOMES:
Number of participants with postoperative complications probably not related to the presence of a patent foramen ovale | First postoperative week
  Complications probably not related to the presence of a patent foramen ovale
Number of days before walking without help | One year
Number of days at home during the first postoperative year | one year
  Number of days of stay at home
Mortality | Three months and one year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - CHU, Rennes